CLINICAL TRIAL: NCT02397954
Title: A Phase 2a Study to Establish the Safety and Tolerability of Zimura™ (Anti-C5 Aptamer) in Combination With Anti-VEGF Therapy in Subjects With Idiopathic Polypoidal Choroidal Vasculopathy (IPCV)
Brief Title: A Study to Establish the Safety and Tolerability of Zimura™ (Anti-C5 Aptamer) in Combination With Anti-VEGF Therapy in Subjects With Idiopathic Polypoidal Choroidal Vasculopathy (IPCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPH2002
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Polypoidal Choroidal Vasculopathy
Keywords: idiopathic polypoidal choroidal vasculopathy; IPCV; Zimura™ (previous name); Avastin®; Eylea®; Lucentis®
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — Bevacizumab; aflibercept; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avacincaptad Pegol + Anti-VEGF (Experimental): Subjects will receive monthly intravitreous injections of Avacincaptad Pegol in combination with either Lucentis, Avastin or Eylea.
  Interventions: Drug: Avacincaptad Pegol

INTERVENTIONS:
Drug: Avacincaptad Pegol — Subjects will receive monthly intravitreous injections of Avacincaptad Pegol in combination with Lucentis, Avastin or Eylea.
  Other Names: Zimura (previous name); IZERVAY; Avastin; Eylea; Lucentis; ARC1905

SUMMARY:
The objectives of this study are to evaluate the safety and tolerability of Zimura™ intravitreous injection in combination with anti-vascular endothelial growth factor (VEGF) therapy in subjects with Idiopathic Polypoidal Choroidal Vasculopathy (IPCV).

DETAILED DESCRIPTION:
Treatment experienced (Prior treatment with anti-VEGF monotherapy of ≥8 injections in the previous twelve (12) months) subjects of either gender aged 50 years or above with a diagnosis of IPCV, will receive 3 monthly (Q4W) intravitreal injections of Zimura™ (1 mg/eye) in combination with anti-VEGF therapy (Avastin® 1.25 mg/eye or Lucentis® 0.5 mg/eye or Eylea® 2 mg/eye).

Safety endpoints include visual acuity loss (proportion of subjects with >15 letter loss at Month 3), ophthalmic adverse events (AEs), systemic adverse events (AEs), change in total retinal thickness (SD-OCT) at Month 3, regression and/or elimination of polyps at Month 3 compared to screening as measured by indocyanine green angiography (ICGA), and laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged ≥ 50 years
* Diagnosis of IPCV
* Treatment-experienced defined as prior treatment with anti-VEGF mono therapy of ≥ 8 injections in the previous twelve (12) months

Exclusion Criteria:

* Any intraocular surgery or thermal laser within three (3) months of trial entry
* Any prior thermal laser in the macular region, regardless of indication
* Any ocular or periocular infection in the twelve (12) weeks prior to entry
* History of any of the following conditions or procedures in the study eye: Rhegmatogenous retinal detachment, pars plana vitrectomy, filtering surgery (e.g. trabeculectomy), glaucoma drainage device, corneal transplant
* Previous therapeutic radiation in the region of the study eye
* A diagnosis of diabetic retinopathy (presence of microaneurysms or any vasculopathy and/or leakage from retinal vasculature in a subject with diabetes mellitus)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2015-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=26397&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Zimura + Anti-VEGF: Zimura 1mg/eye intravitreal injection + Anti-vascular endothelial growth factor (VEGF) (Avastin 1.25mg/eye or Lucentis 0.5mg/eye or Eylea 2mg/eye) intravitreal injection
Period: Overall Study
Arm/Group | Zimura + Anti-VEGF
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Zimura + Anti-VEGF: Zimura 1mg/eye intravitreal injection + Anti-VEGF (Avastin 1.25mg/eye or Lucentis 0.5mg/eye or Eylea 2mg/eye) intravitreal injection
Arm/Group | Zimura + Anti-VEGF
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (6.03)
Age, Customized [Count of Participants; unit: Participants]
  Age: Adults 50-65 | 0
  Age: Adults >65-75 | 2
  Age: Adults >75 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With >15 ETDRS Letter Loss at Month 3
Description: Number of participants with >15 ETDRS letter loss (with calculated percentage)
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Zimura + Anti-VEGF
Number analyzed (Participants) | 4
Participants | 0

2. Primary Outcome: Number of Participants With Ophthalmic Adverse Events
Description: Number of Participants with Ophthalmic Adverse Events (with calculated percentage)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Zimura + Anti-VEGF
Number analyzed (Participants) | 4
Participants | 3

3. Primary Outcome: Number of Participants With Systemic Adverse Events
Description: Number of Participants with Systemic Adverse Events (with calculated percentage)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Zimura + Anti-VEGF
Number analyzed (Participants) | 4
Participants | 1

4. Other Pre Specified Outcome: Mean Change in Central Subfield Retinal Thickness (SD-OCT) From Baseline at Month 3
Description: Mean change in central subfield retinal thickness from baseline at Month 3 as measured by SD-OCT
Time Frame: Baseline and Month 3
Population: Limited sample size; all study participants were included in the analysis.
Measure: Mean (Full Range); unit: μm
Arm/Group | Zimura + Anti-VEGF
Number analyzed (Participants) | 4
μm | -2.75 [-67 to 69]

5. Other Pre Specified Outcome: Regression and/or Elimination of Polyps at Month 3
Description: Regression and/or Elimination of Polyps from baseline to Month 3
Time Frame: Baseline and Month 3
Measure: Number; unit: Polyps
Arm/Group | Zimura + Anti-VEGF
Number analyzed (Participants) | 4
Polyps | NA — Data is not available due to the limited quality of the images

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Zimura + Anti-VEGF
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zimura + Anti-VEGF (N=4)
Endophthalmitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zimura + Anti-VEGF (N=4)
Conjunctival haemorrhage (Eye disorders) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution agrees not to individually publish the results of the Study without Ophthotech's prior written consent. Institution may participate in a joint, multi-center publication of the Study results with other investigators and/or institutions only, upon the prior written consent of Ophthotech.